CLINICAL TRIAL: NCT01417715
Title: Advanced Endoscopic Imaging Using Endomicroscopy for Assessment of Mucosal Healing in IBD
Brief Title: Endomicroscopy for Assessment of Mucosal Healing
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0008
Record Dates: First submitted 2011-08-10; First posted 2011-08-16 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Crohn´s Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Crohn´s disease - active: Patients with Crohn´s disease in the active phase.
  Interventions: Device: Endomicroscopy
- Crohn´s disease - quiescent: Patients with Crohn´s disease in the quiescent phase.
  Interventions: Device: Endomicroscopy
- Ulcerative colitis - active: Patients with ulcerative colitis in the active stage.
  Interventions: Device: Endomicroscopy
- Ucerative colitis - quiescent: Patients with ulcerative colitis in the quiescent stage.
  Interventions: Device: Endomicroscopy

INTERVENTIONS:
Device: Endomicroscopy — Patients will undergo advanced endoscopic imaging using endomicroscopy. Findings will be compared to histopathological and clinical results.

SUMMARY:
Inflammatory bowel disease (IBD) encompasses two major forms of chronic intestinal disorders, Crohn's disease and ulcerative colitis (UC). Diagnosis is based on several macroscopic and histologic features including patterns of inflammation, crypt abscesses and granulomas. Confocal laser endomicroscopy (CLE) is rapidly emerging as a valuable tool for gastrointestinal endoscopic imaging, enabling the endoscopist to obtain an "optical biopsy" of the gastrointestinal mucosa during the endoscopic procedure.

The main objective of this study is to determine endomicroscopic features of mucosal healing in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Residing in institutions (e.g. prison)
* Known allergy against fluorescein
* Proctocolectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn´s disease and ulcerative colitis in the active and quiescent phase of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mucosal healing | up to three years
  We will determine endomicroscopic features of mucosal inflammation (e.g. goblet cell depletion, leackage, microvessel density) in IBD in order to establish a new endoscopic classification of mucosal healing.

SECONDARY OUTCOMES:
Histologic correlation | up to three years
  Comparison of clinical and histopathological data with endoscopic findings to evaluate mucosal healing as a parameter of remission and relapse in patients with IBD.
Therapeutic effect | up to three years
  We will evaluate the effect of different therapeutic strategies (eg. anti-TNF treatment) on characteristics of mucosal healing (e.g. goblet cell depletion, microvessels, leakage).

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Professor, Principal Investigator — Department of Medicine I, University of Erlangen-Nuremberg, Germany; Markus F. Neurath, Professor, Principal Investigator — Department of Medicine I, University of Erlangen-Nuremberg, Germany
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Germany